CLINICAL TRIAL: NCT05322577
Title: A Phase 1b/2 Study Evaluating the Safety, Tolerability, Efficacy, and Pharmacokinetics of Bemarituzumab in Combination With Other Anti-cancer Therapies in Subjects With Previously Untreated Advanced Gastric or Gastroesophageal Junction Cancer (FORTITUDE-103).
Brief Title: A Study Evaluating Bemarituzumab in Combination With Other Anti-cancer Therapies in Subjects With Previously Untreated Advanced Gastric or Gastroesophageal Junction Cancer.
Acronym: FORTITUDE-103
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 20210099
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Cancer
Keywords: Gastric Cancer; Gastroesophageal Junction Cancer; Bemarituzumab; FGFR2b Overexpression
MeSH Terms: conditions — Stomach Neoplasms | interventions — bemarituzumab; Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 Cohort A: Bemarituzumab with CAPOX (Experimental)
  Interventions: Drug: Bemarituzumab; Drug: CAPOX
- Part 1 Cohort C: Bemarituzumab with CAPOX and Nivolumab (Experimental)
  Interventions: Drug: Bemarituzumab; Drug: CAPOX; Drug: Nivolumab
- Part 1 Cohort D: Bemarituzumab with SOX and Nivolumab (Experimental)
  Interventions: Drug: Bemarituzumab; Drug: SOX; Drug: Nivolumab
- Part 2: Bemarituzumab with SOX and Nivolumab. (Experimental)
  Interventions: Drug: Bemarituzumab; Drug: SOX; Drug: Nivolumab

INTERVENTIONS:
Drug: Bemarituzumab — Intravenous (IV) infusion
Drug: CAPOX — CAPOX administered as a combination of oxaliplatin as an IV infusion and capecitabine orally as tablets.
  Arms: Part 1 Cohort A: Bemarituzumab with CAPOX; Part 1 Cohort C: Bemarituzumab with CAPOX and Nivolumab
Drug: SOX — SOX administered as a combination of oxaliplatin as an IV infusion and S-1 orally.
  Arms: Part 1 Cohort D: Bemarituzumab with SOX and Nivolumab; Part 2: Bemarituzumab with SOX and Nivolumab.
Drug: Nivolumab — IV infusion.
  Arms: Part 1 Cohort C: Bemarituzumab with CAPOX and Nivolumab; Part 1 Cohort D: Bemarituzumab with SOX and Nivolumab; Part 2: Bemarituzumab with SOX and Nivolumab.

SUMMARY:
The main objectives of this study are to evaluate the safety and tolerability of bemarituzumab in combination with other anti-cancer therapies, and to evaluate the efficacy of bemarituzumab in combination with S-1 and oxaliplatin (SOX) and nivolumab as assessed by objective response.

ELIGIBILITY:
Inclusion Criteria:

* Adults with unresectable, locally advanced or metastatic gastric or gastroesophageal junction cancer not amendable to curative therapy.
* Ability to provide tumor sample, either archival (obtained within 6 months to joining study) or fresh biopsy.
* For certain arms for Part 1, FGFR2b overexpression positive defined as any FGFR2b 2+/3+ TC determined by centrally performed immunohistochemistry (IHC), based on tumor sample provided.
* For Part 2, FGFR2b overexpression positive defined as FGFR2b ≥10% 2+/3+ TC determined by centrally performed IHC testing, based on tumor sample provided.
* Easter Cooperative Oncology Group (ECOG) performance score less than or equal to 1.
* Measurable or non-measurable disease as long as evaluable by Response Evaluation Criteria Solid Tumors (RECIST) version 1.1
* Participant has no contradictions to CAPOX/SOX plus or minus nivolumab.
* Adequate organ function.
* For Part 2, measurable disease according to RECIST v1.1.

Exclusion Criteria:

* Prior treatment for metastatic or unresectable disease (Note: prior adjuvant or neo-adjuvant therapy for local disease is allowed if ended more than 6 months of 1st dose).
* Prior treatment with any selective inhibitor of fibroblast growth factor - fibroblast growth factor receptor (FGF-FGFR) pathway.
* Known human epidermal growth factor receptor 2 (HER2) positive
* Untreated or symptomatic central nervous system (CNS) disease or brain metastases.
* Peripheral sensory neuropathy greater than or equal to Grade 2.
* Clinically significant cardiac disease.
* Other malignancy within the last 2 years (exceptions for definitively treated disease).
* Chronic or systemic ophthalmological disorders.
* Major surgery or other investigational study within 28 days of first study treatment dose.
* Palliative radiotherapy within 14 days of first study treatment dose.
* Abnormalities of the cornea that may pose an increased risk of developing a corneal ulcer.
* History or evidence of systemic disease or ophthalmological disorders requiring chronic use of ophthalmic corticosteroids.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2026-08-12 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants Who Experience a Dose-limiting Toxicity (DLT) | Day 1 up to Day 21
Part 1: Number of Participants Who Experience a Treatment-emergent Adverse Event (TEAE) | Day 1 to end of treatment (up to approximately 1 year)
Part 2: Objective Response (OR) as per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) | Up to 30 Months

SECONDARY OUTCOMES:
Part 1: Area Under the Concentration-time Curve (AUC) of Bemarituzumab | Day 1 to end of treatment (up to approximately 1 year)
Part 1: Maximum Observed Concentration (Cmax) of Bemarituzumab | Day 1 to end of treatment (up to approximately 1 year))
Part 1: Observed Concentration at the end of a Dose Interval (Ctrough) of Bemarituzumab | Day 1 to end of treatment (up to approximately 1 year)
Part 1: OR per RECIST v1.1 | Up to 2 years
Part 1: Duration of Response (DoR) per RECIST v1.1 | Up to 2 years
Part 1: Disease Control Rate (DCR) | Up to 2 years
Part 1: Progression-free Survival (PFS) per RECIST v1.1 | Up to 2 years
Part 1: Overall Survival (OS) | Up to 2 years
Part 2: Number of Participants Who Experience TEAEs | Up to 30 months
Part 2: DoR per RECIST v1.1 | Up to 30 months
Part 2: Time to Response (TTR) per RECIST v1.1 | Up to 30 months
Part 2: Disease Control (DC) per RECIST v1.1 | Up to 30 months
Part 2: PFS per RECIST v1.1 | Up to 30 months
Part 2: OS | Up to 30 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (42):
- Northport Veterans Affairs Medical Center, Northport, New York, United States
- Japan (31):
  - Fujita Health University Hospital, Toyoake-shi, Aichi-ken
  - Hirosaki University Hospital, Hirosaki-shi, Aomori
  - Chiba University Hospital, Chiba, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Fukui Prefectural Hospital, Fukui-shi, Fukui
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Gifu University Hospital, Gifu, Gifu
  - Ogaki Municipal Hospital, Ogaki-shi, Gifu
  - Gunma University Hospital, Maebashi, Gunma
  - Gunma Prefectural Cancer Center, Ota-shi, Gunma
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima, Hiroshima
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Ibaraki Prefectural Central Hospital, Kasama-shi, Ibaraki
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - St Marianna University Hospital, Kawasaki-shi, Kanagawa
  - Kanagawa Prefectural Hospital Organization Kanagawa Cancer Center, Yokohama, Kanagawa
  - Kochi Health Sciences Center, Kochi, Kochi
  - Kyoto University Hospital, Kyoto, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Okayama University Hospital, Okayama, Okayama-ken
  - Osaka General Medical Center, Osaka, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki-shi, Osaka
  - Shizuoka General Hospital, Shizuoka, Shizuoka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Dokkyo Medical University Hospital, Shimotsuga-gun, Tochigi
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
  - IMSUT Hospital, The Institute of Medical Science The University of Tokyo, Minato-ku, Tokyo
  - Toyama University Hospital, Toyama, Toyama
- National University Hospital, Singapore, Singapore
- South Korea (7):
  - National Cancer Center, Goyang-si Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com